CLINICAL TRIAL: NCT05070559
Title: Comparison of Active Release Technique and Graston Technique In Patients With Chronic Lateral Epicondylitis
Brief Title: Active Release Technique and Graston Technique in Patients With Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Iqra Shabbir
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Lateral Epicondylitis
Keywords: lateral Epicondylitis; Graston Technique; Active Release Technique; Grip Strength
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Release Technique Group (Experimental): Patients in this group will receive Active Release Technique along with conventional therapy
  Interventions: Other: Active Release Technique
- Graston Technique Group (Experimental): Patients in this group will receive Instrumental Assisted Soft Tissue Mobilization along with conventional therapy
  Interventions: Other: Graston Technique Group

INTERVENTIONS:
Other: Active Release Technique — Patients in this group will receive Active Release Technique along with conventional therapy. ART will be given with patient seated, elbow flexed and resting on the treatment table, forearm in midprone & wrist in neutral position and then the therapist will work on the common extensor tendon by applying pressure to the tendon distal to their attachment at the elbow. The patient will start with the elbow bent and wrist straight. As the therapist hold the muscles, the patient will extend the elbow and pronate and flex the wrist while the therapist move the pressure proximally, attempting to release adhesions around and between muscle planes. Total of 15 repetitions for of 10 minutes.
  CONVENTIONAL THERAPY:
  * Hot pack for 15 minutes
  * TENS for 15 minutes
  * Ultrasound (pulsed mode, 1MHz at 1.5 W/cm2 for 5 minutes)
  Arms: Active Release Technique Group
Other: Graston Technique Group — Patients in this group will receive IASTM along with conventional therapy. In graston technique proper application of GT3 which include application of a cream to the common extensor tendon. The GT3will be then used to common extensor tendon. In areas of increased tissue restriction, more required pressure with GT3 is applied using increased force and shorter strokes over the areas of restriction. Ice will be offered as needed for pain management after each session.
  The study includes interventional protocol of 4 weeks. The sessions will be given 3 times a week for 4 weeks.
  CONVENTIONAL THERAPY:
  * Hot pack for 15 minutes
  * TENS for 15 minutes
  * Ultrasound (pulsed mode, 1MHz at 1.5 W/cm2 for 5 minutes)
  Arms: Graston Technique Group

SUMMARY:
This study will be a randomized control trial and will be conducted in Pakistan Railway Hospital Rawalpindi. A sample of 36 participants will be taken. Patients will be divided into two groups by sealed envelop method. Patients in group A will receive Active Release Technique along with conventional therapy while Patients in group B will receive instrument assisted soft tissue mobilization along with conventional therapy. The study includes intervention protocol of 4 weeks. The sessions will be given 3 times a week for 4 weeks. The outcome measures Numeric pain rating scale(NPRS), Hand Dynamometer and Patient-Rated Tennis Elbow Evaluation (PRTEE) will be measured at baseline and at the end of 4th week. Data will be analyzed by SPSS 25

DETAILED DESCRIPTION:
Lateral epicondylitis is an injury caused by overusing the elbow. It is characterized by tenderness and pain over the lateral epicondyle of the elbow. It is not exactly a condition involving inflammation rather a chronic degeneration of the tendon. The major symptom of lateral epicondylitis is presentation or complaint of sharp pain at the lateral side of the elbow with swelling

ELIGIBILITY:
Inclusion Criteria:

* Chronic lateral epicondylitis, complaints for at least 3 months or more
* Pain intensity level between 3 to 6 on 0-10 point numerical pain rating scale

Exclusion Criteria:

* Acute/ sub-acute lateral epicondylitis
* Any cervical spine or any other upper limb dysfunction
* Any other neurological disease, cardiovascular disease, osteoporosis
* Bilateral complaints

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 4 Weeks
  The Numeric Pain Rating Scale that is a unidimensional measure of pain intensity in adults. The 11-point numeric scale ranges from '0' representing one pain extreme (no pain) to '10' representing the other pain extreme (or "worst pain imaginable"). The intrarater reliability with ICC = 0.67.
Hand Dynamometer | 4 Weeks
  hand dynamometer is the most reliable and acceptable tool for measuring grip strength. It detects and quantitatively determines the degree of weak grip strength. (ICC = 0.99)
Patient-Rated Tennis Elbow Evaluation | 4 Weeks
  The Patient-Rated Tennis Elbow Evaluation questionnaire is a specific questionnaire available for assessing the functional status of patients with lateral epicondylitis. (ICC = 0.96)

CONTACTS AND LOCATIONS:
Overall Officials: Sajjad Ali, Ms-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Rawal General Hospital Rawalpindi, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No